CLINICAL TRIAL: NCT02399826
Title: A Prospective, Randomized, Comparative Parallel Study of Amniotic Membrane Graft in the Management of Diabetic Foot Ulcers
Brief Title: Study of Amniotic Membrane Graft in the Management of Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lower Extremity Institute for Research and Therapy (Other)
Collaborators: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Foot; Foot Ulcer; Diabetic
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Other): Surgical debridement of diabetic foot ulcer, followed by collagen alginate and gauze dressing application to be changed daily by patient. Patient will practice offloading, reassessment weekly at office visit
  Interventions: Device: Offloading
- Amniotic Membrane / Amnioband (Experimental): Application of Amnioband with dressing application, to be changed weekly following surgical debridement. Patient will practice offloading. If the ulcer is not closed completely Amnioband will be applied weekly at weeks 2-11
  Interventions: Device: Offloading; Procedure: Dressing Application

INTERVENTIONS:
Device: Offloading — Provision of an offloading cam walker or cast boot, may also convert to "total contact cast" and add felt or foam to supplement
Procedure: Dressing Application — Application of a non adherent dressing, and a multi-layer compression dressing
  Arms: Amniotic Membrane / Amnioband

SUMMARY:
This is comparison trial comparing human amniotic membrane to standard wound care for non healing diabetic foot wounds over a 12 weeks period

DETAILED DESCRIPTION:
This is a prospective, stratified, randomized, comparative, parallel group, Multi-center clinical trial comparing the proportion of ulcers completely healed by use of amniotic membrane graft (Amnioband)versus the standard protocol of wound care in diabetic patients with a diabetic foot ulcer with adequate arterial perfusion, for wound healing to the affected limb. The investigators will compare the proportion of ulcers completely healed by the amniotic membrane graft protocol of care to the standard protocol of care in the management of indolent diabetic ulcers at 6 weeks. In addition the investigators will compare the proportion of healing at 4 weeks, 12 weeks and, the mean time to healing, and the cost effectiveness of the two protocols of care. Mean time to healing will be measured by wound tracings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 18 or older.
2. Patient is willing to provide informed consent and is willing to participate in all procedures and follow up evaluations necessary to complete the study.
3. Patient's ulcer must be diabetic in origin and larger than 1 cm2.
4. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per ADA).
5. Ulcer must be present for a minimum of four weeks before enrollment randomization, with documented failure of conventional ulcer therapy to heal the wound.
6. A two week run-in period will precede enrollment/ randomization in the trial to document the indolent nature of the wounds selected.
7. Additional wounds may be present but not within 3 cm of the study wound.
8. Wound must be present anatomically on the foot as defined by beginning below the malleoli of the ankle and be neuropathic in origin.
9. Patient's ulcer must exhibit no clinical signs of infection.
10. Serum Creatinine less than 3.0mg/dl within last six months.
11. HbA1c less than or equal to 12% within last 90 days.
12. Patient has adequate circulation to the affected extremity, as demonstrated by one of the following within the past 60 days:

    * Dorsum transcutaneous oxygen test (TcPO2) with results ≥30mmHg,
    * ABIs with results of ≥0.7 and ≤1.2, OR
    * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of affected leg

Exclusion Criteria:

1. Patients presenting with an ulcer probing to tendon, muscle, capsule or bone (UT Grade IIIA-D). A positive probe-to-bone will be confirmed when bone or joint can be felt with a sterile, ophthalmological probe.
2. Patients whose index diabetic foot ulcers are greater than 25 cm2.
3. Patients considered not in reasonable metabolic control, confirmed by an HbA1c greater than 12% within previous 90 days.
4. Patients whose serum creatinine levels are 3.0mg/dl or greater within the last six months.
5. Patients with a known history of poor compliance with medical treatments.
6. Patients who have been previously randomized into this study, or are presently participating in another clinical trial.
7. Patients who are currently receiving radiation therapy or chemotherapy.
8. Patients with known or suspected local skin malignancy to the index diabetic ulcer.
9. Patients diagnosed with autoimmune connective tissues diseases.
10. Non-revascularizable surgical sites.
11. Active infection at site.
12. Any pathology that would limit the blood supply and compromise healing.
13. Patients that have received a biomedical or topical growth factor for their wound within the previous 30 days.
14. Patients who are pregnant or breast feeding.
15. Patients who are taking medications that are considered immune system modulators which could affect graft incorporation.
16. Patients with known hypersensitivity to components of any treatment used in the trial.
17. Wounds greater than one year in duration without intermittent healing.
18. Wounds improving greater than 20% over the first two weeks (run-in period) of the trial using standard of care dressing and camboot.
19. Patients taking Cox-2 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of ulcers completely healed by amniotic memrane versus standard care | 6 weeks
  The primary objective of this study is to compare the proportion of ulcers completely healed by the amniotic membrane graft protocol of care to the standard protocol of care in the management of indolent diabetic ulcers at 6 weeks

SECONDARY OUTCOMES:
Proportion of ulcers healed by amniotic membrane versus standard care | 12 weeks
  The secondary objectives of this study are to compare the proportion of healing at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Didomenico, DPM, Principal Investigator — medical director
Locations (3):
- United States (3):
  - Lower Extremity Institute of Research and Therapy, Canfield, Ohio
  - Martinsville Research Institute, Danville, Virginia
  - Shenandoah Lower Extremity Research Institute, Troutville, Virginia